CLINICAL TRIAL: NCT04483271
Title: The Effect of Omega-3 Supplements on the Serum Levels of Selected Cytokines Involved in Cytokine Storm of Covid-19; A Randomized Clinical Trial in the Covid-19 Uninfected Jordanian People
Brief Title: The Effect of Omega-3 on Selected Cytokines Involved in Cytokine Storm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman Abu-Samak, Mahmoud S Abu-Samak, PhD Study Principal Investigator Department of Clinical Pharmacy and Therapeutics, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-PHA-18
Record Dates: First submitted 2020-07-18; First posted 2020-07-23 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cytokine Storm; Cytokines
Keywords: Covid-19; IL-1 beta; IL-6; TNF alpha; Omega-3; n-3FA; uninfected
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3FA group (Experimental): Dietary Supplement: 1,000 mg of wild salmon and fish oil complex once daily, which contains 300 mg of omega3-FA for 2 months.
  Interventions: Dietary Supplement: 300 mg of omega3-FA
- Control group (No Intervention): No intervention was given

INTERVENTIONS:
Dietary Supplement: 300 mg of omega3-FA — The participant will receive 1,000 mg of wild salmon and fish oil complex once daily, which contains 300 mg of omega3-FA.
  Baseline and follow-up serum levels of IL-1,IL-6, and TNF will be measured.
  Other Names: n-3FA
  Arms: n-3FA group

SUMMARY:
The trial was designed to assess the effect of daily dose of 300 mg omega-3 supplements for 2 months on the selected interleukins levels in uninfected people with Covid-19.

DETAILED DESCRIPTION:
Omega-3 Fatty Acids (Omega-3) are long poly unsaturated fatty acids that can be found in plants and fish, its refer to a group composed of three type of fatty acids called: Eicosapentaenoic acid (EPA), Alpha-linoleic acid (ALA), and Docosahexaenoic acid (DHA) . The health promoting effect of n-3FA may be due to immune modulating and anti-inflammatory actions . The anti-inflammatory properties of n-3FA are used for treatment of the inflammatory diseases such as irritable bowel syndrome, rheumatoid arthritis, eczema, and psoriasis . Many studies reported a significant reduction in the risk of cancers in breast, prostate, ovaries with supplementation of n-3FA (Larsson et al. 2004) .However, high-doses omega-3 supplements such as 1000 mg/day are widely spread in community pharmacies in Jordan . Currently , community pharmacy around the world are facing the challenge of increased demand for care of uninfected people with Covid -19. Accordingly , the current randomized clinical trial was designed to evaluate the effect of daily 300 mg of omega 3-FA supplements on the immune health status of uninfected people with Covid-19 as a part of as a part of preventive health care .

Therefore , this RCT aims to assess whether regular daily dose of regular daily dose of omega 3-FA (300 mg) for 2 months supplementation against COVID-19 infection as a part of preventive treatment protocol in uninfected Jordanian peoples. The investigators hypothesize that the regular dose of omega 3-FA (300 mg) /day for 2 months will significantly change immune responses compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included males and females in the age range of 30-66 years without a medical diagnosis of COVID-19 infection.

Exclusion Criteria:

* Exclusion criteria included males or females diagnosed with any chronic immune problems, including autoimmune diseases, chronic or severe infections.
* Pregnant, breastfeeding, and females using hormonal contraceptives were also excluded.

Ages: 30 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
IL-1 beta | (2 months ; 60 days )
  pg/mL
IL-6 | (2 months ; 60 days )
  pg/ml
TNF alpha | (2 months ; 60 days )
  pg/ml

SECONDARY OUTCOMES:
Lipid profile | (2 months ; 60 days )
  mg/dL
Fasting blood glucose | (2 months ; 60 days )
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Study Chair — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan; Rafeef A Al-Khaled, MSC, Principal Investigator — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan
Locations (1):
- Mahmoud S Abu-Samak, Amman, Jordan